CLINICAL TRIAL: NCT06385704
Title: Changes in Intestinal Barrier Function and Gut Microbiome After Duodenal Mucosal Resurfacing
Brief Title: Research on Changes in Intestinal Barrier Function and Gut Microbiome in Patients With Type 2 Diabetes After Duodenal Mucosal Resurfacing (DMR)
Acronym: DMR-IBF-GM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wang Siqi (Other)
Collaborators: China-Japan Friendship Hospital (Other)
Responsible Party: Sponsor-Investigator, Wang Siqi, medical doctor, China-Japan Friendship Hospital
Organization: China-Japan Friendship Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DMRIBFGM0420
Record Dates: First submitted 2024-04-23; First posted 2024-04-26 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; Duodenal Mucosal Resurfacing; Intestinal Barrier Function; Gut Microbiome
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- DMR Procedure (Experimental): Subjects receive the endoscopic DMR procedure in this arm
  Interventions: Procedure: DMR Procedure

INTERVENTIONS:
Procedure: DMR Procedure — Endoscopic procedure

SUMMARY:
The aim of this study is to demonstrate the effects of duodenal mucosal resurfacing (DMR) on intestinal barrier function and gut microbiota when treating uncontrolled type 2 diabetes. Subjects who underwent DMR and those who did not were enrolled, and potential differences were identified by analyzing urine and fecal samples through microbiotic analysis and High Performance Liquid Chromatography (HPLC), combined with changes in clinical data.

DETAILED DESCRIPTION:
This study aims to enroll 100 patients diagnosed with type 2 diabetes who have suboptimal control with one or more oral antidiabetic drugs. Of these, 50 will receive DMR treatment at the Metabolic Weight Loss Center of the China-Japan Friendship Hospital and will be followed up, while the other 50, who have not received DMR treatment, will be matched by age and gender for comparison. Each patient or their legal guardian will sign an informed consent form to participate in the study. Researchers will be granted access to the patients' medical records and will collect their medical history and treatment data. Researchers will also collect urine and fecal samples for microbiome analysis，metagenomics-based studies and HPLC, analyzing the changes in intestinal barrier function and gut microbiota before and after DMR treatment, and between DMR-treated and non-DMR-treated patients.

ELIGIBILITY:
Inclusion Criteria:

- 1.25-65 years of age. 2.Diagnosed with type 2 diabetes. 3.Glycated Hemoglobin (HbA1c) of 7.5 - 10.0% (59-86 mmol/mol). 4.Body Mass Index (BMI) ≥ 24 and ≤ 40 kg/m2. 5.Currently taking one or more oral glucose lowering medications, with no changes in dose or medication in the previous 12 Weeks prior to study entry.

6.Able to comply with study requirements and understand and sign the informed consent.

Exclusion Criteria:

1. Clinical diagnosis of type 1 diabetes.
2. Current use of Glucagon-like peptide-1 (GLP-1) analogues.
3. Hypoglycemia unawareness or a history of severe hypoglycemia.
4. Clinical diagnosis of autoimmune disease.
5. Previous gastrointestinal surgery that could affect the ability to treat the duodenum.
6. Use of anticoagulation therapy (such as warfarin) which cannot be discontinued for 7 days before and 14 days after the procedure.
7. Clinical diagnosis of anemia.
8. Not potential candidates for surgery or general anesthesia.
9. Participating in another ongoing clinical trial of an investigational drug or device.
10. Any other mental or physical condition which, in the opinion of the Investigator, makes the subject a poor candidate for clinical trial participation.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Microbiome Analysis | one week and one month post-treatment
  Characterization of of gut microbiome using next generation sequencing technology
High Performance Liquid Chromatography | one week and one month post-treatment
  Intestinal barrier function using HPLC technology